CLINICAL TRIAL: NCT05945147
Title: Feasibility Study Comparing a Ketamine and Midazolam Infusion to a Midazolam-Only Infusion for Complex Regional Pain Syndrome
Brief Title: Ketamine and Midazolam Infusions for CRPS: Feasibility Study
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Theresa Lii, Principal Investigator, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 66661
Record Dates: First submitted 2023-06-26; First posted 2023-07-14 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Complex Regional Pain Syndromes
Keywords: Feasibility Study; Ketamine; Midazolam; Complex Regional Pain Syndrome; Active Placebo; Analgesics; Dissociative Anesthetics; Chronic Pain; Neuropathic Pain
MeSH Terms: conditions — Complex Regional Pain Syndromes; Chronic Pain; Neuralgia | interventions — Ketamine; Midazolam; Saline Solution; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Ketamine and Midazolam (Experimental): Participants will receive intravenous infusions of ketamine and midazolam for 4 hours each day, over 5 consecutive days, in an outpatient setting.
  Interventions: Drug: Ketamine; Drug: Midazolam
- Midazolam and Saline (Placebo Comparator): Participants will receive intravenous infusions of midazolam and normal saline for 4 hours each day, over 5 consecutive days, in an outpatient setting.
  Interventions: Drug: Midazolam; Drug: Normal Saline

INTERVENTIONS:
Drug: Ketamine — An escalating dose of ketamine (0.15 to 0.4 mg/kg/hr) will be administered as 4-hour infusions over 5 consecutive days
  Other Names: Ketalar
  Arms: Ketamine and Midazolam
Drug: Midazolam — A constant dose of midazolam (0.04 mg/kg/hr) will be administered as 4-hour infusions over 5 consecutive days
  Other Names: Versed
Drug: Normal Saline — An escalating dose of normal saline (0.15 to 0.4 mg/kg/hr) will be administered as 4-hour infusions over 5 consecutive days
  Other Names: 0.9% Sodium Chloride
  Arms: Midazolam and Saline

SUMMARY:
This study will assess the feasibility of administering ketamine plus midazolam or midazolam alone, when infused over 5 days in an outpatient setting, to adults with complex regional pain syndrome (CRPS).

DETAILED DESCRIPTION:
Subanesthetic ketamine infusions are a potentially impactful treatment for chronic refractory pain, but the acute psychoactive effects of ketamine complicate successful masking in randomized trials. Multi-day ketamine infusions have produced long-lasting, but not permanent, remission of symptoms in complex regional pain syndrome (CRPS), a chronic and often debilitating neuropathic pain condition that can affect one or more limbs. In this feasibility study, 4 adults with CRPS will be randomized to receive either ketamine and midazolam or midazolam-only, infused over 5 days in an outpatient setting. The objectives of this feasibility study are:

1. Assess whether the recruitment and retention rate observed in this feasibility study can support a larger clinical trial.
2. Evaluate whether participants can adhere to study procedures.
3. Determine whether midazolam, when given alone as an intravenous (IV) infusion, can be used as an active placebo that is well-tolerated, practical, and believable compared to a ketamine plus midazolam infusion.
4. Gather preliminary data on clinically-relevant outcomes for CRPS.

ELIGIBILITY:
* Age 18 to 65 years
* Meets the International Association for the Study of Pain (IASP) diagnostic criteria for complex regional pain syndrome (CRPS)
* Primary complaint of CRPS-attributable pain for ≥3 months
* Average pain intensity of ≥3/10 over the last month
* Can read and comprehend English-language questionnaires
* Can receive text messages by phone
* Can identify a responsible adult who can provide transportation to and from infusion site for 5 consecutive days (Mon-Fri)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2099-01-01 (Estimated); Primary Completion 2099-04-30 (Estimated); Study Completion 2099-05-31 (Estimated)

PRIMARY OUTCOMES:
Number and proportion of patients who can undergo the steps of recruitment, informed consent, enrollment, and randomization | 2 months after the study opens for enrollment
  Out of all patients identified as potentially eligible for the study based on chart review, we will measure the number and proportion who can undergo the steps of recruitment, informed consent, enrollment, and randomization during a 2-month period.
Number and proportion of randomized participants who remain in the study until the last follow-up timepoint | 8 weeks after receiving intervention
  Out of all patients who were randomized to a treatment group, we will measure the number and proportion who remain in the study until their last follow-up timepoint.
Change in participant masking | Daily during intervention administration (5 days), and once at 8 weeks after receiving intervention
  Participants will be asked to guess their assigned treatment in a forced binary choice and to rate their level of confidence on a scale from 0 to 100%.
Change in participant masking | During intervention administration
  Participants will be asked to guess their assigned treatment in a forced binary choice and to rate their level of confidence on a scale from 0 to 100%.
Change in investigator masking | 8 weeks after receiving intervention
  Investigators administering and monitoring the drug infusions will be asked to guess the participant's assigned treatment in a forced binary choice and to rate their level of confidence on a scale from 0 to 100%.
Change in investigator masking | During intervention administration
  Investigators administering and monitoring the drug infusions will be asked to guess the participant's assigned treatment in a forced binary choice and to rate their level of confidence on a scale from 0 to 100%.
Number and types of adverse events | 8 weeks after receiving intervention
  Adverse events will be elicited from the participant in a brief, open-ended structured interview.

SECONDARY OUTCOMES:
Pain intensity | Baseline, daily during treatment (5 days), and daily for 8 weeks after treatment
  A numerical rating scale ranging from 0 (no pain) to 10 (worst pain imaginable) over the past 24 hours will be used to assess pain intensity.
Treatment expectancies | Baseline, and daily during treatment (5 days)
  The 6-item Healing Encounters and Attitudes Lists (HEAL) Short Form for Treatment Expectancy will be used to assess self-reported expectations about the study treatment. Participants are asked to rate their agreement with brief statements such as, "This treatment will be successful" and "I am confident in this treatment".
Pain interference | Baseline, and weekly for 8 weeks after the end of treatment
  The 6-item PROMIS Pain Interference Short Form assesses the extent to which pain hinders engagement with social, cognitive, emotional, physical, and recreational activities. Items are self-rated on a 5-point scale ranging from 1 ("Not at all") to 5 ("Very Much"). Raw score totals are converted to standardized T-scores, with a higher T-score representing greater pain interference.
Physical function | Baseline, and weekly for 8 weeks after the end of treatment
  The 6-item PROMIS Physical Function Short Form assesses the ability to carry out physical tasks and activities in one's daily life. Items are self-rated on a 5-point scale ranging from 1 ("Unable to do") to 5 ("Without any difficulty"). Raw score totals are converted to standardized T-scores, with a higher T-score representing better physical function.
Depression (PROMIS) | Baseline, and weekly for 8 weeks after the end of treatment
  The 6-item PROMIS Depression Short Form assesses the severity of depressive symptoms experienced by an individual. Items are self-rated on a 5-point scale ranging from 1 ("Never") to 5 ("Always"). Raw score totals are converted to standardized T-scores, with a higher T-score representing greater depression symptom severity.
Depression (PHQ-9) | Baseline, and weekly for 8 weeks after the end of treatment
  The 9-item PHQ-9 will be used as an additional indicator for changes in depression symptom severity, and to monitor for any risk of acute suicidality during the trial (item #9: "Thoughts that you would be better off dead, or of hurting yourself"). Items are self-rated on a 4-point scale ranging from 0 ("Not at all") to 3 ("Nearly every day"). Higher total scores indicate greater depression symptom severity.
Anxiety | Baseline, and weekly for 8 weeks after the end of treatment
  The 6-item PROMIS Anxiety Short Form assesses the severity of anxiety symptoms experienced by an individual. Items are self-rated on a 5-point scale ranging from 1 ("Never") to 5 ("Always"). Raw score totals are converted to standardized T-scores, with a higher T-score representing greater anxiety symptom severity.
Sleep disturbance | Baseline, and weekly for 8 weeks after the end of treatment
  The 6-item PROMIS Sleep Disturbance Short Form assesses the severity of sleep-related issues, such as trouble falling asleep, staying asleep, and experiencing non-restorative sleep. Items are self-rated on a 5-point scale ranging from 1 ("Not at all") to 5 ("Very Much"). Raw score totals are converted to standardized T-scores, with a higher T-score representing greater sleep disturbance.
Pain catastrophizing | Baseline, and weekly for 8 weeks after the end of treatment
  The 13-item Pain Catastrophizing Scale assesses the extent to which an individual engages in magnifying, rumination, and helplessness thoughts related to their pain experience. Items are self-rated on a 5-point scale ranging from 0 ("Not at all") to 4 ("All the time"). Higher total scores indicates higher levels of pain catastrophizing.
Chronic pain acceptance | Baseline, and weekly for 8 weeks after the end of treatment
  The 8-item Chronic Pain Acceptance Questionnaire assesses one's level of acceptance and willingness to engage in valued activities despite the presence of chronic pain. Items are self-rated on a 7-point scale ranging from 0 ("Never true") to 6 ("Always true"). Higher total scores indicate greater levels of chronic pain acceptance.
Patient global impression of change | Weekly for 8 weeks after the end of treatment
  The Patient Global Impression of Change scale assesses the patient's perception of change in their overall health status resulting from a specific treatment. The single-item scale is self-rated on a 7-point scale ranging from 1 ("Very much improved") to 7 ("Very much worse").
Number of painful body regions | Baseline, and weekly for 8 weeks after the end of treatment
  The CHOIR Body Map is a visual tool that allows individuals to indicate the location(s) of their pain on a human body outline.

CONTACTS AND LOCATIONS:
Overall Officials: Theresa R Lii, MD, MS, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No